CLINICAL TRIAL: NCT02415231
Title: "The Effect of Humor and Laughter on C Reactive Protein: A Pilot Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gurinder Bains, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5150100
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: humor laughter C reactive protein
MeSH Terms: interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- humor (Experimental): humor group will watch humor video for 20 minutes
  Interventions: Behavioral: humor
- control non humor (No Intervention): control group did not watch humor, they sat quietly for 20 minutes.

INTERVENTIONS:
Behavioral: humor
  Arms: humor

SUMMARY:
The study is to see if watching humor and laughing can affect CRP levels in healthy individuals. This is a randomized controlled trial.

DETAILED DESCRIPTION:
Subjects will be…males and females: students, employees, and members of the community.

5. "Subjects will be between ___18_ and ___99_ years of age."

6. "In total, subject participation will last approximately ___1 day for 90 minutes_

7. "Subjects will be recruited _by word of mouth at the Loma Linda University Campus and surrounding communities___."

8. "Consent will take place _by investigators in Nichol Hall Room A620/A640___."

9. If Multi-center:

10. If Single center or investigator-initiated:

"_60__ subjects will participate in the study."

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-99 yrs , healthy individuals

Exclusion Criteria:

* Under 18 years old, or over 99 years old, non healthy individuals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
CRP level | change in CRP levels over 3 time frames (baseine, immediately after intervention, and 30 minutes later)

CONTACTS AND LOCATIONS:
Overall Officials: gurinder bains, MD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Nichol Hall Room A640, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No